CLINICAL TRIAL: NCT03291847
Title: Maternal Buprenorphine-naloxone Treatment During the Perinatal Period: Fetal and Infant Effects
Brief Title: Maternal Buprenorphine-naloxone Treatment and the Infant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00093171; 1R01DA041367-01A1 (NIH)
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Maternal Opioid Use Disorder; Opioid Exposed Infant
Keywords: maternal opioid use; neonatal abstinence syndrome; buprenorphine-naloxone
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Fetal Monitoring; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: A group of n=40 study participants will receive buprenorphine-naloxone medication assisted therapy for the treatment of opioid use disorder during pregnancy. This group will undergo fetal monitoring at 24, 28, 32 and 36 weeks of gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Buprenorphine-naloxone treated (Experimental): Participants receiving buprenorphine-naloxone treatment for opioid use disorder during pregnancy
  Interventions: Device: fetal monitoring; Drug: Buprenorphine Naloxone

INTERVENTIONS:
Device: fetal monitoring — Maternal fetal monitoring
  Other Names: maternal physiology monitoring
Drug: Buprenorphine Naloxone — Treatment for opioid use disorder
  Other Names: Suboxone

SUMMARY:
The purpose of this mechanistic study is to evaluate the effects that maternal buprenorphine-naloxone maintenance have on the neurobehavioral development of the fetus and infant. To accomplish this, the investigators will study a sample of 120 opioid dependent pregnant women that will receive buprenorphine-naloxone as part of substance abuse treatment at a comprehensive care treatment facility for pregnant and parenting women with substance use disorders. Fetal neurobehavior and maternal physiology will be assessed, via an established maternal-fetal data acquisition system, at 4 points during gestation: 24, 28, 32 and 36 weeks. Infant birth parameters and Neonatal Abstinence Syndrome (NAS) spectrum display will be evaluated at birth, and infant neurodevelopment will be assessed during the first month of life.

DETAILED DESCRIPTION:
The project population will be 40 pregnant women with opioid use disorder inducted as outpatients to buprenorphine-naloxone maintenance. Subject treatment data, including medical and obstetric histories, drug use histories, demographic information and psychosocial information will be extracted from patient charts. Weekly urine toxicology testing will provide information regarding other substance use/misuse during the time of study participation. Study participants will undergo 2 60 minute maternal and fetal neurophysiologic monitoring sessions on one day at 4 points during gestation: 24, 28, 32 and 36 weeks, at times of trough (just before sublingual buprenorphine-naloxone or methadone daily dose) and peak (2 1/2 hours after dosing) maternal drug levels. Fetal cardiac (heart rate, heart rate variability, heart rate accelerations) and movement (total fetal movement, number and duration of movement bouts) and the correlation between the two (fetal heart rate-movement coupling) will be determined. Maternal physiologic measures will include heart period and variability, vagal tone, skin conductance and respiratory data. All maternal and fetal measures, with the exception of blood pressure, will be computed in 1-minute intervals and averaged over the 60 min recording. Infant birth data and birth parameters, and neonatal abstinence syndrome scores will be extracted from patient charts. Infants will undergo neurobehavioral testing using the Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale, a 30 minute harmless assessment of infant functioning, on days 3, 14 and 30 of life.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid use disorder (OUD) as defined by DSM V criteria
* singleton pregnancies, generally uncomplicated by conditions that jeopardize pregnancy outcome
* Gestation less than 24 weeks

Exclusion Criteria:

* Complications of pregnancy, including gestational diabetes, polyhydramnios, hypertension, placenta previa or significant risk of preterm delivery;
* Evidence of fetal malformation detected by prenatal ultrasound;
* Significant general maternal health problems that can affect fetal functioning, including Type I or gestational diabetes, alterations in thyroid functioning, HIV infection or hypertension;
* Significant maternal psychopathology that would preclude informed consent;
* Alcohol use disorder per DSM V criteria (see ascertainment methods below)
* Women stable on methadone maintenance (defined as more than 3 consecutive days of dosing)
* Women coming to treatment reporting "street" methadone use (for more than 3 consecutive days
* Women not planning to receive obstetric care at the Center for Addiction and Pregnancy; - Women not planning to deliver their infants at Johns Hopkins Bayview Medical center
* Women planning for adoption of their infant.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women with opioid use disorder
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine-naloxone Treated
Started | 42
Completed (There were 26 fetuses associated with 24 women) | 24
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: Data not collected for subjects removed from the study
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate at 24 Weeks
Description: Fetal heart rate in beats per minute, mean over 60 minutes gestation. Fetal heart rate in msec at 24 weeks of gestation at times of peak maternal plasma drug concentrations
Time Frame: 24 weeks of gestation
Population: Fetal monitoring performed for all participants enrolled in the study at that gestational age who met criteria for monitoring
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 13
Number analyzed (Fetuses) | 13
beats per minute | 143.64 (4.38)

2. Primary Outcome: Fetal Heart Rate at 28 Weeks Gestation
Description: Fetal heart rate in beats per minute, mean over 60 minutes gestation. Fetal heart rate at 28 weeks of gestation at times of tpeak maternal plasma drug concentrations.
Time Frame: 28 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 16
Number analyzed (Fetuses) | 16
beats per minute | 139.14 (3.93)

3. Primary Outcome: Fetal Heart Rate at 32 Weeks Gestation
Description: Fetal heart rate in beats per minute, mean over 60 minutes. Fetal heart rate at 32 weeks of gestation at times of peak maternal plasma drug concentrations
Time Frame: 32 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 19
Number analyzed (Fetuses) | 19
beats per minute | 135.82 (146.83)

4. Primary Outcome: Fetal Heart Rate at 36 Weeks Gestation
Description: Fetal heart rate in beats per minute, mean over 60 minutes. Fetal heart rate at 36 weeks of gestation at times of peak maternal plasma drug concentrations.
Time Frame: 36 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 15
Number analyzed (Fetuses) | 15
beats per minute | 131.99 (5.52)

5. Primary Outcome: Total Fetal Movement at 24 Weeks Gestation
Description: Total fetal movement at 24 weeks of gestation. Total number of fetal moves over 60 minutes via fetal monitoring at time of peak maternal plasma drug concentrations at 24 weeks of gestation.
Time Frame: 24 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fetal movements
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 11
Number analyzed (Fetuses) | 11
fetal movements | 71.91 (13.8)

6. Primary Outcome: Total Fetal Movement at 36 Weeks Gestation
Description: Total fetal movement over 60 minutes via fetal monitoring at 36 weeks of gestation. Nimber of fetal movements over 60 minutes via fetal monitoring at times of peak maternal plasma drug concentrations at 36 weeks of gestation.
Time Frame: 36 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fetal movements
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 15
Number analyzed (Fetuses) | 15
fetal movements | 59.07 (17.17)

7. Primary Outcome: Total Fetal Movement at 28 Weeks Gestation
Description: Total fetal movement over 60 minutes via fetal monitoring. Total fetal movement over 60 minutes via fetal monitoring at times of trough and peak maternal plasma drug concentrations at 28 weeks of gestation.
Time Frame: 28 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fetal movements
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 15
Number analyzed (Fetuses) | 15
fetal movements | 70.06 (12.13)

8. Primary Outcome: Total Fetal Movement at 32 Weeks Gestation
Description: Total fetal movement over 60 minutes via fetal monitoring at 32 weeks of gestation. Number of fetal moves over 60 minutes via fetal monitoring at times of peak maternal plasma drug concentrations at 32 weeks of gestation.
Time Frame: 32 weeks of gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fetal movements
Units Other Than Participants: Fetuses
Arm/Group | Buprenorphine-naloxone Treated
Number analyzed (Participants) | 18
Number analyzed (Fetuses) | 18
fetal movements | 66.00 (19.13)

ADVERSE EVENTS:
Time Frame: From the time of protocol enrollment up to 30 days of infant age, an average of 6 months
Description: Any adverse pregnancy or neonatal complication was reported. All pregnancies were tracked via the project obstetrician from the time of study enrollment until delivery. All infants were tracked from the time of delivery through 30 days of age.
  There were 26 pregnancies during the study. Two women had two pregnancies each.
Arm/Group | Buprenorphine-naloxone Treated
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 3/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine-naloxone Treated (N=26)
pectus carinatum, mild (Musculoskeletal and connective tissue disorders) | 1 (1) — Also low set ears. Determined to be morphologically similar to the father of the baby.
missed spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Subject was inducted onto study medication at 11 weeks of gestation; she miscarried at fetus sized 7 weeks 6 days 3 days later. It was determined that the subject was not viably pregnant at the time of study medication induction
congenital malformation (Gastrointestinal disorders) | 1 (1) — Infant was born with mild CHARGE association (presumed); most likely unrelated to study medication

LIMITATIONS AND CAVEATS:
The COVID pandemic greatly affected the program from which participants were drawn and thereby subject enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03291847/Prot_SAP_000.pdf